CLINICAL TRIAL: NCT03630640
Title: Immunotherapy by Nivolumab in Neoadjuvant and Adjuvant Setting in Patients With Advanced HCC Treated by Electroporation in Curative Intent: French Multicenter Phase 2 Therapeutic Trial.
Brief Title: Neoadjuvant and Adjuvant Nivolumab in HCC Patients Treated by Electroporation
Acronym: NIVOLEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P171001J
Record Dates: First submitted 2018-07-09; First posted 2018-08-15 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: nivolumab; neoadjuvant; electroporation,adjuvant
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Electroporation

STUDY DESIGN:
Intervention Model Description: Clinical study phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab Injection [Opdivo] (Experimental): Intravenous Nivolumab 240 Q2W neoadjuvant Intravenous Nivolumab 480 mg Q4W- adjuvant for 12 months
  Interventions: Drug: Nivolumab Injection [Opdivo]

INTERVENTIONS:
Drug: Nivolumab Injection [Opdivo] — Intravenous Nivolumab 240 Q2W neoadjuvant Intravenous Nivolumab 480 mg Q4W- adjuvant up to 12 months after EP
  Other Names: Irreversible electroporation

SUMMARY:
Percutaneous ablation (PA) is the only non-surgical curative treatment of hepatocellular carcinoma (HCC). Due to its excellent tolerance, particularly in patients with portal hypertension or bearing comorbidities, it now represents in France nearly 70% of the first-line curative treatment of "in Milan" tumours. For HCC less than 3 cm, ideal indication for percutaneous ablations, results of monopolar radiofrequency ablation (mRFA), are excellent with only 5% of reported non-tumoral control after a first procedure .

In addition to mRFA the arsenal of ablations has grown considerably with the emergence of new techniques. They allow the expansion of indications for PA, especially in patients with poor prognostic tumors or relatively advanced beyond the Milan criteria . In this setting, multibipolar mode using no touch technique (mbpRFAnt) increases the tumour volume that can be ablated, allowing the removal of large tumors> 5 cm . Furthermore, electroporation (EP) is a new PA technique that does not promote thermoablation but induce tumoral cells apoptosis and is particularly interesting for difficult-to-treat lesions located near vascular or biliary trunks . Inadequate tumour control is then de facto greater in these situations, around 20% at one year.

The idea of optimizing HCC curative treatments using neoadjuvant or adjuvant biotherapy, particularly in patients with advanced tumors in curative intent, is particularly attractive. One trial in adjuvant setting was conducted, the STORM trial, that tested the benefit of sorafenib in curative intent of in Milan HCC. This negative trial included patients with in Milan HCC, with an expected low rate of recurrence with only few patients treated by PA.

In parallel, the development of new molecules for HCC treatment, especially immunotherapy, seems to give promising results in palliative setting . Furthermore, PA procedures and most likely electroporation induce T-cell recruitement that may foster immunomodulation .

Neoadjuvant and adjuvant trials using these new molecules must now be cautiously designed based on the rigorous selection of special populations and therapeutic indications.

This project proposes a Phase 2 trial testing the safety and efficacy of treatment with Nivolumab in neoadjuvant and adjuvant setting in patients with advanced HCC treated by electroporation in curative intent.

DETAILED DESCRIPTION:
Multicenter (6 centers), Phase 2 trial.

-Inclusion visit The inclusion visit takes place between 15 days and no later than 3 days before the patient's hospitalization for Neoadjuvant therapy

Eligible patients will receive :

* 2 nivolumab infusions in a neoadjuvant setting (every 15 days) The treatment will be carried out every 2 weeks s, for 2 cycles before EP procedure The patient is hospitalized one day for treatment
* EP procedure performed in a curative attempt EP procedure will be performed according to previously described procedure in the setting of routine management of HCC as decided in multidisciplinary boards in each centre.
* 12 nivolumab infusions in an adjuvant setting (every 30 days) during one year. The patient is hospitalized one day for infusion
* Classical follow-up during an additional year (every 3 months) Follow up after adjuvant therapy (M12-M24) The usual evaluation will be performed every 3 months

Constitution of a biobank with :

* paraffin and frozen tumoral and non tumoral biopsy sampled at before and after one month of neoadjuvant Nivolumab (second biopsies at the time of the electroporation procedure)
* Serum samples and Peripheral blood mononuclear cells (PBMC) before and after one month of neoadjuvant Nivolumab then after EP at 1, 3, 6, 9 and 12 months after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Histological diagnosis of HCC, whether new or recurrent following a prior curative therapeutic management > 6 months.
* Barcelona Clinical Liver Cancer(BCLC) stage Category A
* Patients with HCC eligible for EP as assessed by multidisciplinary board corresponding to the following extension:

  * Uninodular HCC≥ 2 cm and ≤ 5 cm, no macroscopic vascular invasion
  * Multinodular HCC maximum 3 nodules ≤ 3 cm, no macroscopic vascular invasion
* At least one uni-dimensional measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to modified RECIST for HCC
* Liver function status Child-Pugh Class A
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Adequate bone marrow, liver and renal function
* Life expectancy ≥ 3 months
* Women of childbearing potential and men must agree to use adequate contraception
* Patients affiliated to a Social Security System
* Written informed consent signed

Exclusion Criteria:

* Patients with contraindications to EP (Pacemakers or patients who have a history of cardiac arrhythmias or irregular heartbeats, ascites, Coagulopathy, Ongoing infection)
* Patients with contraindication to contrast medium intravenous injection either gadolinium or iodinate
* Prior liver transplantation or candidates for liver transplantation
* Prior systemic treatment for HCC, in particular agents targeting T-cell costimulation or checkpoint pathways (including those targeting PD-1, PD-L1 or PD-L2, CD137, or cytotoxic T-lymphocyte antigen [CTLA-4]).
* Patients with uncontrolled HBV infection and viral load above 100 IU/mL.
* Patients with large esophageal varices at risk of bleeding that are not being treated with conventional medical intervention
* Past or concurrent history of neoplasm other than HCC, except for in situ carcinoma of the cervix uteri and/or non-melanoma skin cancer and superficial bladder tumors. Any cancer curatively treated > 3 years prior to study entry is permitted
* Known history or symptomatic metastatic brain or meningeal tumors
* Major surgical procedure or significant traumatic injury within 28 days before enrolment
* Congestive heart failure New York Heart Association (NYHA) ≥ class 2
* Unstable angina or myocardial infarction within the past 6 months before enrolment
* Grade 3 (severe) hypertension ≥180 and/or ≥110 mmHG (systolic and diastolic, according to National Heart Foundation 2016)
* Patients with phaeochromocytoma
* Refractory ascites according to EASL guidelines definition (ascites that cannot be mobilized or the early recurrence of which cannot be prevented because of a lack of response to sodium restriction and diuretic treatment)
* Persistent proteinuria of NCI-CTCAE version 4.0 ≥ Grade 3
* Ongoing infection > Grade 2 according to NCI-CTCAE version 4.0. Hepatitis B is allowed if no active replication is present (HBV replication below 100 IU/mL). Hepatitis C is allowed if no antiviral treatment is required
* Clinically significant bleeding NCI-CTCAE version 4.0 ≥ Grade 3 within 30 days before enrolment
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident, deep vein thrombosis or pulmonary embolism within 6 months before enrolment
* Any psychological, familial, sociological, geographical or illness or medical condition that could jeopardize the safety of the patient and/or his compliance with the study protocol and follow-up procedure
* Known history of human immunodeficiency virus (HIV) infection
* Seizure disorder requiring medication
* Non-healing wound, ulcer or bone fracture
* Known hypersensitivity to the study drug or excipients in the formulation
* Any malabsorption condition
* Breast feeding
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-08-19 (Actual)

PRIMARY OUTCOMES:
Local recurrence-free survival during a 1-year follow-up after Nivolumab neoadjuvant/adjuvant therapy and EP procedure | At 1 year
  Recurrence rates (whether local or distant) will be assessed using imaging techniques as recommended by international guidelines (3-months US and MRI during two years). Patients who will meet primary endpoint will be alive 1 year after EP procedure without evidence of local recurrence on 3-months US/MRI evaluations.

SECONDARY OUTCOMES:
Changes of tumorous and non-tumorous perfusion parameters observed with CUS and MRI after one months of neoadjuvant treatments | after one month of neoadjuvant treatment
  Evaluation performed by CUS and MRI
Per nodule rates of early response | At one month after a single procedure of EP
  Evaluation performed by MRI
Incidences of intra segmental/ extra segmental distant recurrence | During follow-up (2 yrs)
  Evaluation performed by MRI
Assessment of overall survival | At 2-yrs following EP procedure
  patients will meet this endpoint if they are alive with or without HCC recurrence 2 years after EP. procedures. Causes and date of death will be specified when applicable during this timeframe.
Assessment of tolerance of the immunotherapy treatment: | During follow-up (2 yrs)
  Adverse events related to Nivolumab infusions will be monitored according to manufacturer guidelines and recommendation.
Compliance to neoadjuvant treatments | During follow-up (13 months)
  Respect of scheduled Nivolumab infusions
Compliance to adjuvant treatments | During follow-up (13 months)
  Respect of scheduled Nivolumab infusions
Frequency of SAEs | During follow-up (2 yrs)
  adverse events related to Nivolumab infusions will be monitored according to manufacturer guidelines and recommendation.
Frequency of discontinuations treatment due to AEs | During follow-up (2 yrs)
  adverse events related to Nivolumab infusions will be monitored according to manufacturer guidelines and recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre NAHON, MD,PhD, Principal Investigator — APHP-Hôpital Jean Verdier
Locations (1):
- Hôpital Jean Verdier, Bondy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutter O, Calvo J, N'Kontchou G, Nault JC, Ourabia R, Nahon P, Ganne-Carrie N, Bourcier V, Zentar N, Bouhafs F, Sellier N, Diallo A, Seror O. Safety and Efficacy of Irreversible Electroporation for the Treatment of Hepatocellular Carcinoma Not Amenable to Thermal Ablation Techniques: A Retrospective Single-Center Case Series. Radiology. 2017 Sep;284(3):877-886. doi: 10.1148/radiol.2017161413. Epub 2017 Apr 28. PMID 28453431
- [Background] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648